CLINICAL TRIAL: NCT00003849
Title: A Phase II Trial of C2B8 in Patients With Asymptomatic CD20+ B-Cell Follicular Small Cleaved Low-Grade Non-Hodgkin's Lymphoma or Relapsed CD20+ Hodgkin's Disease
Brief Title: Rituximab in Treating Patients With Non-Hodgkin's Lymphoma or Hodgkin's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-987851; NCI-2012-02298 (Registry Identifier: CTRP (Clinical Trials Reporting System)); CDR0000067010 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 1999-11-01; First posted 2004-05-03 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-07

CONDITIONS: Lymphoma
Keywords: recurrent adult Hodgkin lymphoma; stage III grade 1 follicular lymphoma; stage IV grade 1 follicular lymphoma
MeSH Terms: conditions — Lymphoma; Hodgkin Disease; Lymphoma, Follicular | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- rituximab (Experimental): Patients receive rituximab IV over 4-6 hours on day 1 weekly for 4 weeks. Patients are followed at 1, 3, 6, 9, and 12 months, then every 6 months for 3 years, then annually thereafter.
  Interventions: Biological: rituximab

INTERVENTIONS:
Biological: rituximab

SUMMARY:
RATIONALE: Monoclonal antibodies can locate cancer cells and either kill them or deliver cancer-killing substances to them.

PURPOSE: Phase II trial to study the effectiveness of rituximab in treating patients who have non-Hodgkin's lymphoma or Hodgkin's disease.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the response rate (complete or partial) to rituximab in previously untreated patients with stage III or IV CD20+ B-cell follicular small cleaved cell non-Hodgkin's lymphoma. II. Determine the response rate (complete or partial) to rituximab in patients with relapsed CD20+ Hodgkin's disease. III. Determine the time to progression and time to chemotherapy in these patients after treatment with rituximab.

OUTLINE: Patients are stratified according to disease (follicular small cleaved cell non-Hodgkin's lymphoma vs relapsed Hodgkin's disease). Patients receive rituximab IV over 4-6 hours on day 1 weekly for 4 weeks. Patients are followed at 1, 3, 6, 9, and 12 months, then every 6 months for 3 years, then annually thereafter.

PROJECTED ACCRUAL: A total of 21-32 patients will be accrued for each arm of this study within 7-10.5 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven stage IIIA or stage IVA B-cell follicular small cleaved cell non-Hodgkin's lymphoma Tumor cells express CD20 No prior chemotherapy or radiotherapy Stable disease that would otherwise be observed OR Histologically proven relapsed Hodgkin's disease of any stage Tumor cells express CD20 Bidimensionally measurable disease Masses (e.g., enlarged lymph nodes) must be at least 1.5 cm X 1.5 cm by CT, MRI, or x-ray Splenic enlargement considered measurable if spleen palpable at least 3 cm below the left costal margin No CNS lymphoma

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: Not specified Hematopoietic: No more than 5,000 circulating tumor cells Hepatic: Not specified Renal: Not specified Other: Not pregnant or nursing Fertile patients must use effective contraception during and for at least 12 months following study HIV negative No other active malignancies

PRIOR CONCURRENT THERAPY: See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 1999-07; Primary Completion 2005-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
response rate | Up to 5 years

SECONDARY OUTCOMES:
time to progression | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Thomas E. Witzig, MD, Study Chair — Mayo Clinic
Locations (21):
- United States (20):
  - CCOP - Scottsdale Oncology Program, Scottsdale, Arizona
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - Siouxland Hematology-Oncology, Sioux City, Iowa
  - CCOP - Wichita, Wichita, Kansas
  - CCOP - Ochsner, New Orleans, Louisiana
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - CCOP - Duluth, Duluth, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Clinic, Saint Cloud, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Quain & Ramstad Clinic, P.C., Bismarck, North Dakota
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - Altru Health Systems, Grand Forks, North Dakota
  - CCOP - Toledo Community Hospital Oncology Program, Toledo, Ohio
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota
- Saskatchewan Cancer Agency, Regina, Saskatchewan, Canada

REFERENCES:
- [Result] Witzig TE, Vukov AM, Habermann TM, Geyer S, Kurtin PJ, Friedenberg WR, White WL, Chalchal HI, Flynn PJ, Fitch TR, Welker DA. Rituximab therapy for patients with newly diagnosed, advanced-stage, follicular grade I non-Hodgkin's lymphoma: a phase II trial in the North Central Cancer Treatment Group. J Clin Oncol. 2005 Feb 20;23(6):1103-8. doi: 10.1200/JCO.2005.12.052. Epub 2005 Jan 18. PMID 15657404